CLINICAL TRIAL: NCT02884076
Title: Validating the Ability of the Sodergren Score to Guide Management of Symptomatic Haemorrhoids in a Malaysian Population
Brief Title: Validation of Sodergren Score for Haemorrhoids in Malaysia
Status: Completed | Type: Observational
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Galen Sha, Dr, University of Malaya
Other Study IDs: Sodergren Validation
Record Dates: First submitted 2016-08-22; First posted 2016-08-30 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Sodergren score; Validation
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic Hemorrhoid: Consecutive patients with symptomatic hemorrhoids presenting to our clinic

SUMMARY:
To validate the ability of the Sodergren score in guiding the management of symptomatic haemorrhoids in a Malaysian population.

DETAILED DESCRIPTION:
All participating, consented subjects will be scored with the Sodergren score prior to receiving a standardized ambulatory treatment regime. The questionnaire will be self-administered by the subjects. Subjects whom are not able to self-administer the questionnaire will be assisted by the investigator or research assistant. The nature and severity of the subject's haemorrhoidal symptoms are considered as the pre-treatment baseline. A follow up period of 12 months will be carried out post treatment for failure or success of treatment. The data collected will be compared to pre-treatment scores and analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Male and female genders
* Previous ambulatory treatment
* Internal Haemorrhoids

Exclusion Criteria:

* Presence of external haemorrhoids
* Prior haemorrhoidal surgery
* Anti-coagulant therapy
* Anal fissure
* Inflammatory bowel disease
* Underlying colon-rectal malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients at specialist clinics
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Method of treatment | 12 months
  Surgery or ambulatory treatment of hemorrhoid

CONTACTS AND LOCATIONS:
Overall Officials: Hon Leong Sha, MD, Principal Investigator — University of Malaya
Locations (1):
- HRPB, Ipoh, Perak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pucher PH, Qurashi M, Howell AM, Faiz O, Ziprin P, Darzi A, Sodergren MH. Development and validation of a symptom-based severity score for haemorrhoidal disease: the Sodergren score. Colorectal Dis. 2015 Jul;17(7):612-8. doi: 10.1111/codi.12903. PMID 25603811